CLINICAL TRIAL: NCT01982604
Title: A Phase 1, Open-label, Randomized, Crossover Clinical Trial to Evaluate PK/PD of 30 U TI Inhalation Powders Prepared With Insulin From Two Different Suppliers
Brief Title: Comparison of 30 Units of TI (Technosphere® Insulin) Prepared With Insulin From Two Different Suppliers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-179
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence (Group) 1 (Experimental): Subjects randomized to Sequence 1 will receive TI in the following sequence:
  TI-Inhalation Powder A TI-Inhalation Powder B
  *30 units (10 units + 20 units)
  Interventions: Drug: TI-Inhalation Powder A; Drug: TI-Inhalation Powder B
- Sequence (Group) 2 (Experimental): Subjects randomized to Sequence 2 will receive TI in the following sequence:
  TI-Inhalation Powder B TI-Inhalation Powder A
  *30 units (10 units + 20 units)
  Interventions: Drug: TI-Inhalation Powder A; Drug: TI-Inhalation Powder B

INTERVENTIONS:
Drug: TI-Inhalation Powder A — Inhaled Insulin
Drug: TI-Inhalation Powder B — Inhaled Insulin

SUMMARY:
A Phase 1, open-label randomized crossover trial in Healthy Volunteers to evaluate the PK/PD of TI (Technosphere® Insulin) prepared with insulin from two different suppliers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 55 years, considered healthy based on screening physical examination, medical history, clinical chemistry, and urinalysis

  * HNVs with a screening blood pressure less than 140/90 mm Hg
  * Subjects who have hypertension controlled with up to 1 medication and who have a blood pressure less than 140/90 mm Hg
  * Note: For subjects with blood pressure at or above 140/90 mm Hg; two additional readings 5 minutes apart are allowed but the last blood pressure reading must be in range
  * Subjects who have hypercholesterolemia controlled with up to 1 medication and who have a low-density lipoprotein value less than 160 mg/dL
* Good venous access for blood draws
* No smoking in the past 6 months (including cigarettes, cigars, and pipes) and urine cotinine testing < 100 ng/mL
* Body mass index (BMI) < 32 kg/m2
* Completion of informed consent form

Exclusion Criteria:

* Blood donation (500 mL) within the last 8 weeks
* Fasting blood sugar >100 mg/dL
* History of coronary artery disease, peripheral vascular disease, or congestive heart failure
* Allergy to study drug, components of Boost and Boost Plus, or other study material
* Clinically significant active or chronic illness
* History of asthma, COPD, or any other clinically relevant chronic lung disease
* Respiratory tract infection within 4 weeks before screening
* History of drug or alcohol abuse within the past 5 years
* Positive urine drug screen
* Clinically significant screening ECG, physical examination, laboratory test, or vital sign abnormality
* Exposure to any other investigational drug or device within 30 days before treatment or within 90 days before treatment for drugs known to modify glucose metabolism
* History of malignancy within the 5 years before screening (other than basal cell carcinoma)
* History of human immunodeficiency virus (HIV) infection or hepatitis B or C
* Women who are pregnant, lactating, or planning to become pregnant during the clinical study period
* Women of childbearing potential (premenopausal who have not undergone hysterectomy or bilateral tubal ligation, or postmenopausal for fewer than 2 years) not practicing adequate birth control. Adequate birth control is defined as using oral, percutaneous, or transdermal contraceptives; condoms and diaphragms (double barrier) with a spermicide; or intrauterine devices. Postmenopausal for the purposes of this clinical study includes experiencing amenorrhea for 2 or more years or being surgically sterile.
* Any subject who, in the opinion of the PI or a designee, appears not to be qualified for this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
AUC (area-under-the-serum-insulin concentration time curve) 0 - 240 minutes | 5, 10, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 210, 240
Cmax (maximum serum insulin concentration) | 5, 10, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 210, 240

SECONDARY OUTCOMES:
GIR (area-under-the-serum Glucose Infusion Rate) | 0 to 360

CONTACTS AND LOCATIONS:
Locations (1):
- Chula Vista, California, United States